CLINICAL TRIAL: NCT01631890
Title: Phase III Study of the Efficacy of Endoscopic Ultrasound (EUS) Assisted Endoscopic Glue Injection and Conventional Endoscopic Injection Therapy for Prevention of Gastric Variceal Rebleed
Brief Title: To Compare the Efficacy of Endoscopic Ultrasound Assisted Endoscopic Glue Injection and Conventional Endoscopic Injection Therapy for Prevention of Gastric Variceal Rebleed
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILBS- EUS-001
Record Dates: First submitted 2012-06-14; First posted 2012-06-29 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2012-06

CONDITIONS: Bleeding Gastric Varices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard endotherapy (Active Comparator)
  Interventions: Procedure: Standard Endotherapy
- Endoscopic Ultrasound assisted endoscopic glue injection (Experimental)
  Interventions: Procedure: Endoscopic Ultrasound assisted endoscopic glue injection

INTERVENTIONS:
Procedure: Endoscopic Ultrasound assisted endoscopic glue injection — N Butyl cyanoacrylate will be used for achieving initial hemostasis during active gastric variceal bleed and during follow up gastric variceal obturation. Endoscopic injection will be performed intravariceally using a therapeutic endoscope and a steel hubbed catheter, with N-butyl-2-cyanoacrylate. The cyanoacrylate will be injected without dilution with lipiodol. The tip of the endoscope will be coated with lipiodol to prevent sticking of glue to the endoscope. The injection catheter is primed with saline solution followed by injection of glue in 1ml aliquot to fill the dead space followed by injection of sterile water to flush the glue into the varix. The needle is withdrawn immediately after the glue injection to prevent tissue adherence.
  Arms: Endoscopic Ultrasound assisted endoscopic glue injection
Procedure: Standard Endotherapy — Patients will be stabilized by giving i/v fluids, blood and blood products. Injection terlipressin will be given to all patients in a bolus dose of 2mg within 30 minutes of admission to the hospital. This would be followed by 1mg i/v 6hrly and will be continued for 5 days. If terlipressin cannot given then inj.somatostatin 500mcg IV bolus followed by 250mcg/hr continuous infusion for 5days.
  Arms: standard endotherapy

SUMMARY:
Consecutive patients who meet the eligibility criteria will be enrolled into the study. All patients with gastric varices with no history of gastric variceal bleed (Group C) will undergo Endoscopic ultrasound and Upper Gastrointestinal Endoscopy at baseline, at the end of first year and at the end of study.

The patients who presented to Institute of Liver and Biliary Sciences with gastric variceal bleed or develop Gastric Variceal bleed during hospital stay will be randomized into Group -A (conventional Upper Gastrointestinal Endoscopy + Glue) and Group-B (Endoscopic Ultrasound followed by Upper Gastrointestinal Endoscopy+Glue) therapy for gastric varices. Total 90 patients will be enrolled and randomized into group A and Group B after resuscitation and urgent Upper Gastrointestinal Endoscopy with standard therapy for bleeding gastric varices to achieve hemostasis.

ELIGIBILITY:
Inclusion Criteria:

* A clinical, radiological or histologic diagnosis of cirrhosis
* Upper Gastrointestinal endoscopy showing gastric varices
* Informed consent to participate in the study

Exclusion Criteria:

* Previous endotherapy (Endoscopic Variceal Ligation/Esophageal Variceal Sclerotherapy/Endoscopic Variceal Obliteration) for gastric variceal haemorrhage
* Diagnosed case of HepatoPulmonary Syndrome.
* Non -cirrhotic portal hypertension/Extra hepatic Portal Venous Obstruction
* transhepatic intrajugular portosystemic shunt, (balloon-occluded retrograde transvenous obliteration), balloon-occluded endoscopic injection sclerotherapy, shunt operation.
* Hepatic encephalopathy grade III/IV,
* Cardio respiratory failure
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Proportions of patients with gastric varices develops rebleed after complete gastric varices obturation in 2 years | 2 years

SECONDARY OUTCOMES:
Proportion of patients who will achieve complete Gastric variceal obliteration in both groups | 2 years
Proportions of patients who will show adverse effects of gastric variceal obturation by N Butyl cyanoacrylate. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Kr Choudhury, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India